CLINICAL TRIAL: NCT00928473
Title: The Danish Childhood Obesity Biobank
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zealand University Hospital (Other)
Collaborators: University of Copenhagen (Other); Steno Diabetes Center Copenhagen (Other); Holbaek Sygehus (Other)
Responsible Party: Principal Investigator, Jens Christian Holm, MD, PhD, University of Copenhagen
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 250609
Record Dates: First submitted 2009-06-25; First posted 2009-06-26 (Estimated); Last update posted 2020-11-12 (Actual); Status verified 2020-11

CONDITIONS: Obesity; Metabolic Disease; NAFLD, Non-alcoholic Fatty Liver Disease; Cardiovascular Diseases
MeSH Terms: conditions — Obesity; Metabolic Diseases; Non-alcoholic Fatty Liver Disease; Cardiovascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Lifestyle counseling (Experimental): The obese children will start a treatment for obesity in the Children's Obesity Clinic. This treatment includes lifestyle counseling, objective examination, weight-controls, visiting a psychologist, visiting a dietician and blood samples, DXA-scan, eventually MRI.
  Interventions: Behavioral: A family-centered, multidisciplinary obesity treatment program

INTERVENTIONS:
Behavioral: A family-centered, multidisciplinary obesity treatment program — The obese children will start a treatment for obesity in the Children's Obesity Clinic. This treatment includes lifestyle counseling, objective examination, weight-controls, visiting a psychologist, visiting a dietician and blood samples, DXA-scan, eventually MRI.
  Other Names: (Holm, J. C. et al. Chronic care treatment of obese children and adolescents. Int. J. Pediatr. Obes. 6, 188-196, 2011).

SUMMARY:
The Danish Childhood Obesity Biobank aims to produce a scientific platform for research in obesity: Bio-clinical data are collected from two cohorts - an obesity clinic cohort and a population-based cohort. The biobank thus facilitates translation between research and clinical practice of obesity treatment and related complications.

DETAILED DESCRIPTION:
The Danish Childhood Obesity Biobank collects data from two cohorts - an obesity clinic cohort and a population-based cohort, of which the latter functions as a reference group.

The biobank continuously and longitudinally includes clinical data and biological samples from children and adolescents in obesity treatment. The population-based cohort has been recruited in a cross-sectional manner from Danish schools, high schools, and dentistries.

Data included in the biobank include venous blood samples, stool, urine, saliva, anthropometrics, body composition by dual-energy X-ray absorptiometry, magnetic resonance imaging and spectroscopy, and genetic markers among others. The data are stored in a central secured electronic database and biological materials are stored in -80-degree Celsius freezers until analyses.

To date, the Danish Childhood Obesity Biobank have included data from more than 5250 children, adolescents and adults from the obesity clinic cohort and more than 4200 from the population-based cohort.

ELIGIBILITY:
Inclusion Criteria:

* 2- 100 Years old
* Adipose, BMI > 90 % percentile

Ages: 2 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 5000 (Estimated)
Dates: Start 2009-01; Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Weightloss, changes in blood parameters and in fatty liver developement. | continuously

CONTACTS AND LOCATIONS:
Overall Officials: Jens-Christian Holm, Ph.d., MD, Study Chair — The Children's Obesity Clinic and The Danish Childhood Obesity Biobank
Locations (1):
- The Children's Obesity Clinic, Paediatric department, University Hospital Holbæk, Region Zealand, Holbæk, Denmark

REFERENCES:
- [Derived] Stinson SE, Jonsson AE, Andersen MK, Lund MAV, Holm LA, Fonvig CE, Huang Y, Stankevic E, Juel HB, Angquist L, Sorensen TIA, Ongstad EL, Gaddipati R, Grimsby J, Rhodes CJ, Pedersen O, Christiansen M, Holm JC, Hansen T. High Plasma Levels of Soluble Lectin-like Oxidized Low-Density Lipoprotein Receptor-1 Are Associated With Inflammation and Cardiometabolic Risk Profiles in Pediatric Overweight and Obesity. J Am Heart Assoc. 2023 Feb 7;12(3):e8145. doi: 10.1161/JAHA.122.027042. Epub 2023 Jan 25. PMID 36695299
- [Derived] Johansen MJ, Vonsild Lund MA, Angquist L, Fonvig CE, Holm LA, Chabanova E, Thomsen HS, Hansen T, Holm JC. Possible prediction of obesity-related liver disease in children and adolescents using indices of body composition. Pediatr Obes. 2022 Oct;17(10):e12947. doi: 10.1111/ijpo.12947. Epub 2022 Jun 21. PMID 35726748
- [Derived] Frithioff-Bojsoe C, Lund MAV, Lausten-Thomsen U, Fonvig CE, Lankjaer IOJ, Hansen T, Hansen T, Baker JL, Holm JC. Early detection of childhood overweight and related complications in a Danish population-based cohort aged 2-8 years. Obes Res Clin Pract. 2022 May-Jun;16(3):228-234. doi: 10.1016/j.orcp.2022.04.001. Epub 2022 May 3. PMID 35514021
- [Derived] Stinson SE, Jonsson AE, de Retana Alzola IF, Lund MAV, Frithioff-Bojsoe C, Aas Holm L, Fonvig CE, Pedersen O, Angquist L, Sorensen TIA, Holst JJ, Christiansen M, Holm JC, Hartmann B, Hansen T. Hyperglucagonemia in Pediatric Adiposity Associates With Cardiometabolic Risk Factors but Not Hyperglycemia. J Clin Endocrinol Metab. 2022 May 17;107(6):1569-1576. doi: 10.1210/clinem/dgac108. PMID 35213713
- [Derived] Stinson SE, Jonsson AE, Lund MAV, Frithioff-Bojsoe C, Aas Holm L, Pedersen O, Angquist L, Sorensen TIA, Holst JJ, Christiansen M, Holm JC, Hartmann B, Hansen T. Fasting Plasma GLP-1 Is Associated With Overweight/Obesity and Cardiometabolic Risk Factors in Children and Adolescents. J Clin Endocrinol Metab. 2021 May 13;106(6):1718-1727. doi: 10.1210/clinem/dgab098. PMID 33596309
- [Derived] Lund MAV, Thostrup AH, Frithioff-Bojsoe C, Lausten-Thomsen U, Hedley PL, Pedersen O, Christiansen M, Hansen T, Holm JC. Low-grade inflammation independently associates with cardiometabolic risk in children with overweight/obesity. Nutr Metab Cardiovasc Dis. 2020 Aug 28;30(9):1544-1553. doi: 10.1016/j.numecd.2020.04.024. Epub 2020 May 5. PMID 32571613
- [Derived] Jors A, Lund MAV, Jespersen T, Hansen T, Poulsen HE, Holm JC. Urinary markers of nucleic acid oxidation increase with age, obesity and insulin resistance in Danish children and adolescents. Free Radic Biol Med. 2020 Aug 1;155:81-86. doi: 10.1016/j.freeradbiomed.2020.05.009. Epub 2020 May 25. PMID 32464183
- [Derived] Frithioff-Bojsoe C, Lund MAV, Lausten-Thomsen U, Hedley PL, Pedersen O, Christiansen M, Baker JL, Hansen T, Holm JC. Leptin, adiponectin, and their ratio as markers of insulin resistance and cardiometabolic risk in childhood obesity. Pediatr Diabetes. 2020 Mar;21(2):194-202. doi: 10.1111/pedi.12964. Epub 2019 Dec 26. PMID 31845423
- [Derived] Johansen MJ, Gade J, Stender S, Frithioff-Bojsoe C, Lund MAV, Chabanova E, Thomsen HS, Pedersen O, Fonvig CE, Hansen T, Holm JC. The Effect of Overweight and Obesity on Liver Biochemical Markers in Children and Adolescents. J Clin Endocrinol Metab. 2020 Feb 1;105(2):dgz010. doi: 10.1210/clinem/dgz010. PMID 31617910
- [Derived] Viitasalo A, Schnurr TM, Pitkanen N, Hollensted M, Nielsen TRH, Pahkala K, Atalay M, Lind MV, Heikkinen S, Frithioff-Bojsoe C, Fonvig CE, Grarup N, Kahonen M, Carrasquilla GD, Larnkjaer A, Pedersen O, Michaelsen KF, Lakka TA, Holm JC, Lehtimaki T, Raitakari O, Hansen T, Kilpelainen TO. Abdominal adiposity and cardiometabolic risk factors in children and adolescents: a Mendelian randomization analysis. Am J Clin Nutr. 2019 Nov 1;110(5):1079-1087. doi: 10.1093/ajcn/nqz187. PMID 31504107
- [Derived] Hollensted M, Fogh M, Schnurr TM, Kloppenborg JT, Have CT, Ruest Haarmark Nielsen T, Rask J, Asp Vonsild Lund M, Frithioff-Bojsoe C, Ostergaard Johansen M, Vincent Rosenbaum Appel E, Mahendran Y, Grarup N, Kadarmideen HN, Pedersen O, Holm JC, Hansen T. Genetic Susceptibility for Childhood BMI has no Impact on Weight Loss Following Lifestyle Intervention in Danish Children. Obesity (Silver Spring). 2018 Dec;26(12):1915-1922. doi: 10.1002/oby.22308. PMID 30460774
- [Derived] Fonvig CE, Hamann SA, Nielsen TRH, Johansen MO, Gronbaek HN, Mollerup PM, Holm JC. Subjective evaluation of psychosocial well-being in children and youths with overweight or obesity: the impact of multidisciplinary obesity treatment. Qual Life Res. 2017 Dec;26(12):3279-3288. doi: 10.1007/s11136-017-1667-5. Epub 2017 Jul 31. PMID 28762099
- [Derived] Nielsen TRH, Lausten-Thomsen U, Fonvig CE, Bojsoe C, Pedersen L, Bratholm PS, Hansen T, Pedersen O, Holm JC. Dyslipidemia and reference values for fasting plasma lipid concentrations in Danish/North-European White children and adolescents. BMC Pediatr. 2017 Apr 28;17(1):116. doi: 10.1186/s12887-017-0868-y. PMID 28454530
- [Derived] Rischel HE, Nielsen LA, Gamborg M, Moller P, Holm JC. Comparison of sensory-specific satiety between normal weight and overweight children. Appetite. 2016 Dec 1;107:486-493. doi: 10.1016/j.appet.2016.08.123. Epub 2016 Sep 1. PMID 27593452
- [Derived] Trier C, Dahl M, Stjernholm T, Nielsen TR, Bojsoe C, Fonvig CE, Pedersen O, Hansen T, Holm JC. Effects of a Family-Based Childhood Obesity Treatment Program on Parental Weight Status. PLoS One. 2016 Aug 25;11(8):e0161921. doi: 10.1371/journal.pone.0161921. eCollection 2016. PMID 27560141
- [Derived] Fonvig CE, Chabanova E, Ohrt JD, Nielsen LA, Pedersen O, Hansen T, Thomsen HS, Holm JC. Multidisciplinary care of obese children and adolescents for one year reduces ectopic fat content in liver and skeletal muscle. BMC Pediatr. 2015 Dec 30;15:196. doi: 10.1186/s12887-015-0513-6. PMID 26714769
- [Derived] Lausten-Thomsen U, Christiansen M, Fonvig CE, Trier C, Pedersen O, Hansen T, Holm JC. Reference values for serum total adiponectin in healthy non-obese children and adolescents. Clin Chim Acta. 2015 Oct 23;450:11-4. doi: 10.1016/j.cca.2015.07.012. Epub 2015 Jul 10. PMID 26169157
- [Derived] Hvidt KN, Olsen MH, Ibsen H, Holm JC. Weight reduction and aortic stiffness in obese children and adolescents: a 1-year follow-up study. J Hum Hypertens. 2015 Sep;29(9):535-40. doi: 10.1038/jhh.2014.127. Epub 2015 Jan 15. PMID 25589213
- [Derived] Hvidt KN, Olsen MH, Ibsen H, Holm JC. Effect of changes in BMI and waist circumference on ambulatory blood pressure in obese children and adolescents. J Hypertens. 2014 Jul;32(7):1470-7; discussion 1477. doi: 10.1097/HJH.0000000000000188. PMID 24733029
- [Derived] Hvidt KN, Olsen MH, Holm JC, Ibsen H. Obese children and adolescents have elevated nighttime blood pressure independent of insulin resistance and arterial stiffness. Am J Hypertens. 2014 Nov;27(11):1408-15. doi: 10.1093/ajh/hpu055. Epub 2014 Apr 9. PMID 24717420
- [Derived] Lausten-Thomsen U, Nielsen TR, Thagaard IN, Larsen T, Holm JC. Neonatal anthropometrics and body composition in obese children investigated by dual energy X-ray absorptiometry. Eur J Pediatr. 2014 May;173(5):623-7. doi: 10.1007/s00431-013-2226-x. Epub 2013 Dec 7. PMID 24318487
- [Derived] Holm JC, Gamborg M, Neland M, Ward L, Gammeltoft S, Heitmann BL, Sorensen TI, Ibsen KK. Longitudinal changes in blood pressure during weight loss and regain of weight in obese boys and girls. J Hypertens. 2012 Feb;30(2):368-74. doi: 10.1097/HJH.0b013e32834e4a87. PMID 22157326